CLINICAL TRIAL: NCT00150397
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Six-Week Study Of The Efficacy And Safety Of Tofimilast Dry Powder For Inhalation In Adults With Persistent Asthma
Brief Title: A Study of the Safety and Efficacy of Tofimilast in Adult Asthmatics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2641021
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — tofimilast

INTERVENTIONS:
Drug: Tofimilast

SUMMARY:
This is an initial proof of concept, phase to study to assess the safety and efficacy tofimilast for the chronic maintenance treatment of adults with persistent asthma

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate persistent asthma (NAEPP/GINA Step 2-3)
* Reversibility to albuterol at least 12% and 200 mL

Exclusion Criteria:

* Any significant co-morbid disease, particularly cardiovascular
* Use of any maintenance therapy except short acting bronchodilators
* Smoking history > or = 10 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112
Dates: Start 2005-03; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FEV1 compared to placebo

SECONDARY OUTCOMES:
Change from baseline in other lung function parameters, disease control and quality of life compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (16):
  - Pfizer Investigational Site, Encinitas, California
  - Pfizer Investigational Site, Riverside, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Normal, Illinois
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Skillman, New Jersey
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Madison, Wisconsin
- Costa Rica (2):
  - Pfizer Investigational Site, Barrio Aranjuez, Provincia de San José
  - Pfizer Investigational Site, San José, Provincia de San José
- India (4):
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Vellore, Tamil Nadu
  - Pfizer Investigational Site, Noida, Uttar Pradesh

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2641021&StudyName=A+Phase+2+Study+of+the+Safety+and+Efficacy+of+Tofimilast+in+Adult+Asthmatics